CLINICAL TRIAL: NCT06367998
Title: The Effect of Pregabalin on Shoulder Pain of Patients With Myofascial Pain Syndrome and Central Sensitization Who Undergo Arthroscopic Rotator Cuff Repair
Brief Title: Effect of Pregabalin on Shoulder Pain in Patients With Central Sensitization After Arthroscopic Rotator Cuff Repair
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Collaborators: Viatris Korea (Industry)
Responsible Party: Principal Investigator, Hyungsuk Kim, Assistant professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PC24MISV0017
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Rotator Cuff Tears; Central Sensitisation; Neuropathic Pain
MeSH Terms: conditions — Rotator Cuff Injuries; Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin group (Experimental)
  Interventions: Drug: Pregabalin
- Control group (No Intervention)

INTERVENTIONS:
Drug: Pregabalin — Pregabalin oral intake from the day before surgery to six weeks postoperatively
  Other Names: Lyrica
  Arms: Pregabalin group

SUMMARY:
This study aims to investigate the effects of Pregabalin intake on shoulder pain management in patients with central sensitization undergoing arthroscopic rotator cuff repair. Although Pregabalin is known to be effective in controlling pain after shoulder arthroscopy, research on its efficacy in pain management for patients with central sensitization is scarce. Utilizing a list that identifies central sensitization, this study will explore whether Pregabalin can reduce postoperative pain in these patients and potentially improve joint mobility, emotional, and physical functioning. A prospective randomized study is planned, with inclusion criteria set for patients aged between 19 and 70 who have undergone arthroscopic rotator cuff repair.

The study will compare clinical outcomes up to one year postoperatively between two groups of 38 patients each. The case group will receive standard postoperative medications (NSAIDs) plus Pregabalin oral intake from the day before surgery to six weeks postoperatively, while the control group will receive only the standard postoperative medications without Pregabalin.

ELIGIBILITY:
Inclusion Criteria:

* Age over 19 to under 70
* Underwent arthroscopic rotator cuff repair due to a tear of the rotator cuff.
* Clinical diagnosis of myofascial pain syndrome
* Central sensitization (Central Sensitization Inventory (CSI) score of 40 or above).

Exclusion Criteria:

* Previous history of Pregabalin prescription
* Hypersensitivity reactions or severe complications after taking Pregabalin.
* Diagnosed with and are being treated for psychiatric disorders
* Localized infection, sepsis, or previous neurological abnormalities
* Uncontrolled hypertension (evidenced by a resting blood pressure of more than 100 mmHg)
* Liver function abnormalities (aspartate aminotransferase or alanine aminotransferase >60 IU/litre).
* major cardiovascular diseases or renal impairments

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
The Visual Analogue Scale (VAS) pain score | Preoperative, postoperative 2, 6 weeks, 2, 4, 6 and 12 months
  Pain score evaluation from 0 to 10, 10 meaning the maximum pain

SECONDARY OUTCOMES:
Constant shoulder score | Preoperative, postoperative 6 months and 12 months
  Shoulder functional score from 0 to 100, 100 meaning excellent shoulder function
American shouler and elbow surgeons (ASES) score | Preoperative, postoperative 6 months and 12 months
  Shoulder functional score from 0 to 100, 100 meaning excellent shoulder function